CLINICAL TRIAL: NCT02287792
Title: Effect of 18-FDG PET/CT Imaging on Clinical Decision Making During the Acute Phase of Infective Endocarditis: a Multicenter Prospective Impact Study
Brief Title: 18-FDG PET/CT Imaging and Clinical Decisions in Infective Endocarditis
Acronym: TEPvENDO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AOM13549
Record Dates: First submitted 2014-10-31; First posted 2014-11-11 (Estimated); Last update posted 2025-08-08 (Actual); Status verified 2017-07

CONDITIONS: Infective Endocarditis
Keywords: Infective endocarditis; 18-FDG PET/CT; Impact; Patient's management; Diagnostic
MeSH Terms: conditions — Endocarditis; Tooth, Impacted; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | US Export: No

ARMS (1):
- 18-FDG PET/CT scan (Experimental): All patients will undergo a whole body PET/CT scan
  Interventions: Procedure: 18-FDG PET/CT scan

INTERVENTIONS:
Procedure: 18-FDG PET/CT scan — Whole body 18-FDG PET/CT to assess cardiac and extracardiac complications in infective endocarditis

SUMMARY:
The purpose of this study is to assess the impact of 18-FDG positron emission tomography (PET)/computed tomography (CT) imaging in the management of patients with suspected or proven IE in detecting cardiac valve damages and other extracardiac complications. The study will evaluate whether this procedure can change the clinical decisions (treatments, valve surgery, patients' overall care) and modify the diagnosis of IE.

DETAILED DESCRIPTION:
Introduction:

Infective endocarditis (IE) is a rare disease, often difficult to diagnose with a high mortality rate. Extra-cardiac manifestations, which can occur in 30 to 80% of cases, impact the outcome of the disease. Identifying these manifestations may help confirm an uncertain diagnosis and optimize patients' management.

18-FDG PET/CT imaging, widely used for cancer staging, may also detect hyper-metabolic areas related to extracardiac infectious complications of IE. It provides the opportunity to detect all extracardiac IE infectious complications through a single examination. The impact of 18-FDG PET/CT imaging on the management of IE has yet to be completely evaluated.

Hypothesis:

18-FDG PET/CT implementation could result in both shortening of the initial diagnostic work-up of IE and therapeutic optimization.

Primary objective:

To evaluate the impact of 18-FDG PET/CT on patients' management, as measured by changes in IE therapeutic plans.

Secondary objectives:

* To evaluate the impact of 18-FDG PET/CT on the Duke-Li criteria for IE diagnosis
* To evaluate the performance of 18-FDG PET/CT in detecting valve damages and extracardiac complications induced by the IE
* To evaluate whether 18-FDG PET/CT may help identify the infection's portal of entry
* To evaluate whether the detection of extracardiac complications by FDG PET/CT is associated with the 6-months survival rate
* To identify clinical and biological determinants of extracardiac IE localizations and prognosis
* To determine the inter-reader interpretation of the18-FDG PET/CT results and the reproducibility in preparation and acquisition method

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged ≥ 18 years
2. Presenting IE "Duke-Li definite - Duke-Li possible" or strong suspicion of IE "Duke-Li not definite or possible, with initiation of IE antibiotic therapy".
3. Transthoracic or transesophageal ultrasound performed.
4. A stable clinical condition which does not require immediate surgery or contraindicate patient mobilization
5. Absence of cardiac surgery for the current IE episode
6. Covered by the French health insurance system
7. Having given and signed the written study informed consent to the study.

Exclusion Criteria:

1. Patient having already had a 18-FDG PET/CT in the current episode
2. Contraindication to perform a 18-FDG PET/CT
3. Early prosthetic valve IE (cardiac surgery within last 2 months)
4. Inability to understand the information form
5. Pregnant or lactating woman.
6. Cardiac surgery between inclusion and 18-FDG PET/CT
7. Participation to any clinical trial including 18-FDG PET/CT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2015-04-17 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with a change in IE therapeutic plan | 7 days
  at least one modification in antimicrobial or anticoagulant therapy (types, route, dose, number, duration, indication…) or any modification of surgery (type, timing, indications…)

SECONDARY OUTCOMES:
Proportion of patients with Duke-Li classification modifications | 6 months
  Proportion of patients with change in diagnostic classification of IE (definite, possible, excluded) according to the Duke-Li classification
Performances of 18-FDG PET/CT in detection of IE localization as compared to other usual procedures | 6 months
  1/ in detecting valve damages and extracardiac complications and 2/ in identify the portal of entry of IE
6-month mortality rate | 6 months
  number of dead patients 6 months after inclusion
Determinants of change in therapeutic plan as defined in primary outcome | 6 months
  Clinical and biological determinants of therapeutic changes
18-FDG PET/CT inter-reader reproducibility | 6 months
  questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Duval, Professor, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Bichat Claude Bernard Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Boursier C, Duval X, Bourdon A, Imbert L, Mahida B, Chevalier E, Claudin M, Hoen B, Goehringer F, Selton-Suty C, Roch V, Lamiral Z, Humbert O, Rouzet F, Marie PY; AEPEI-TEPvENDO study group. ECG-Gated Cardiac FDG PET Acquisitions Significantly Improve Detectability of Infective Endocarditis. JACC Cardiovasc Imaging. 2020 Dec;13(12):2691-2693. doi: 10.1016/j.jcmg.2020.06.036. Epub 2020 Aug 19. No abstract available. PMID 32828775
- [Background] Duval X, Le Moing V, Tubiana S, Esposito-Farese M, Ilic-Habensus E, Leclercq F, Bourdon A, Goehringer F, Selton-Suty C, Chevalier E, Boutoille D, Piriou N, Le Tourneau T, Chirouze C, Seronde MF, Morel O, Piroth L, Eicher JC, Humbert O, Revest M, Thebault E, Devillers A, Delahaye F, Boibieux A, Gregoire B, Hoen B, Laouenan C, Iung B, Rouzet F; AEPEI-TEPvENDO study group. Impact of Systematic Whole-body 18F-Fluorodeoxyglucose PET/CT on the Management of Patients Suspected of Infective Endocarditis: The Prospective Multicenter TEPvENDO Study. Clin Infect Dis. 2021 Aug 2;73(3):393-403. doi: 10.1093/cid/ciaa666. PMID 32488236
- [Background] Boursier C, Duval X, Mahida B, Hoen B, Goehringer F, Selton-Suty C, Chevalier E, Roch V, Lamiral Z, Bourdon A, Piriou N, Pallardy A, Morel O, Rouzet F, Marie PY; AEPEI-TEPvENDO Study Group. Hypermetabolism of the spleen or bone marrow is an additional albeit indirect sign of infective endocarditis at FDG-PET. J Nucl Cardiol. 2021 Dec;28(6):2533-2542. doi: 10.1007/s12350-020-02050-2. Epub 2020 Feb 10. PMID 32043240